CLINICAL TRIAL: NCT02621879
Title: Bilateral Gluteal Fascio-myo-cutaneous Advancement Flap in Treatment of Recurrent Sacrococcygeal Pilonidal Disease
Brief Title: Bilateral Gluteal Fascio-myo-cutaneous Flap in Treatment of Recurrent Pilonidal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of general surgery, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mansourau27
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bilateral Gluteal Advancement Flap (Experimental): Advancement of both gluteal muscles to the midline after release incisions in their fascia.
  Interventions: Procedure: Bilateral Gluteal Advancement Flap

INTERVENTIONS:
Procedure: Bilateral Gluteal Advancement Flap — Dissection of both gluteus maximus muscles from their origin in the sacrum, advancement of both muscles is conducted to the midline after creating release incisions in their fascia.

SUMMARY:
Bilateral Gluteal Fascio-myo-cutaneous Advancement Flap is a modified technique used in Treatment of Recurrent Sacrococcygeal Pilonidal sinus

DETAILED DESCRIPTION:
Patients with recurrent pilonidal sinus disease are recruited to undergo Bilateral Gluteal Fascio-myo-cutaneous Advancement Flap technique under spinal anesthesia in order to prevent recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent sacrococcygeal pilonidal disease aging more than 16 years with single or multiple pits were included in the study.
* Patients included presented with recurrence of pilonidal disease at least six months after the first operation.

Exclusion Criteria:

* Patients aging less than 16 years.
* Patients unfit for anesthesia.
* Patients with primary pilonidal disease.
* Patients with acute pilonidal abscess or active infection.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Incidence of recurrence | 18 months
  Number of patients who presents with recurrent pilonidal sinus within the follow up period

SECONDARY OUTCOMES:
Incidence of complications | 18 months
  Number of patients who present with wound infection or other morbidity after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, M.D, Principal Investigator — Mansoura Univesity
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided